CLINICAL TRIAL: NCT02576067
Title: Cardiovascular Inflammation Reduction Trial (CIRT) - Inflammation Imaging Study
Brief Title: Cardiovascular Inflammation Reduction Trial - Inflammation Imaging Study
Acronym: CIRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Unity Health Toronto (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Zahi Fayad, Director Translational and Molecular Imaging Institute, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-1382; 1R01HL128056-01A1 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Vascular Inflammation; Atherosclerotic Cardiovascular Disease
Keywords: Atherosclerotic cardiovascular disease; Inflammation reduction
MeSH Terms: conditions — Atherosclerosis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose methotrexate (Experimental): average dose of 15-20 mg po/weekly
  Interventions: Drug: Low dose methotrexate
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose methotrexate — Study participants will additionally receive 1 mg daily oral folate.
  Arms: Low dose methotrexate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Vascular inflammation, a central feature of atherosclerosis, participates in the initiation, perpetuation and instability of plaques. Multiple clinical trials of cholesterol lowering therapy with statins have demonstrated that reductions in atherosclerotic cardiovascular disease (CVD) events are associated with reductions in both LDL cholesterol (LDL-C) and the systemic inflammatory mediator C-reactive protein (CRP). The Cardiovascular Inflammation Reduction Trial (CIRT) investigates if an anti-inflammatory agent commonly used in rheumatoid arthritis (low dose methotrexate (LDM)) can reduce CV morbidity and mortality among patients with a prior myocardial infarction or angiographically demonstrated multivessel coronary artery disease (GCO#13-1467).

In this ancillary CIRT imaging study, the investigators propose to use this well validated approach by non-invasive serial FDG-PET/CT imaging in a subset of patients enrolled in the main CIRT trial to directly visualize vascular inflammation. Once the subjects are enrolled in the main CIRT trial, baseline imaging will be done and follow up imaging will be done approximately 8 months after the baseline imaging.

18FDG-PET imaging data will be acquired, analyzed centrally and results incorporated into the main CIRT database. The investigators hypothesize that LDM treatment will result in a significant decrease in plaque inflammation as measured by 18-FDG-PET/CT after 8 months as compared to placebo.

DETAILED DESCRIPTION:
The NHLBI funded (Ridker 5U01HL101422) Cardiovascular Inflammation Reduction Trial (CIRT) provides a unique opportunity to investigate whether a commonly used anti-inflammatory agent used in rheumatoid arthritis (low dose methotrexate (LDM)) can reduce CVD morbidity and mortality among patients with stable coronary artery disease. CIRT, is a randomized, double-blind, placebo-controlled, multi-center trial among 7,000 men and women with prior myocardial infarction or angiographically demonstrated multivessel coronary artery disease. Eligible participants will be randomly allocated over a three to four year period to usual care plus placebo or usual care plus LDM (average dose of 15-20 mg po/weekly. CIRT proposes that the reduction in CVD events with methotrexate derives from its effect on vascular inflammation, thus it is crucial to incorporate a measure of vascular inflammation imaging for confirmation of the primary mechanism of action underlying CIRT. As such, the direct evaluation of arterial inflammation would enhance the scientific value of the CIRT trial.

The inclusion of the proposed vascular inflammation imaging substudy has widespread implications that will allow this imaging modality to serve as a surrogate measure of disease, and thereby provide an opportunity for stratification in individuals at risk for CVD and evaluation of other interventions with presumed anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at screening
* Documented MI in the past or past evidence of multivessel coronary artery disease by angiography must have completed any planned coronary revascularization procedures associated with the qualifying event, and must be clinically stable for at least 60 d before screening; the qualifying prior MI must be documented either by hospital records or by evidence on current electrocardiogram of Q waves in 2 contiguous leads and/or an imaging test demonstrating wall motion abnormality or scar; the qualifying documentation of multivessel coronary disease must include angiographic evidence of atherosclerosis in at least 2 major epicardial vessels defined either as the presence of a stent, a coronary bypass graft, or an angiographic lesion of 60% or greater. Left main coronary artery disease that has been revascularized with a stent or bypass graft will qualify as multivessel disease, as will the presence of a 50% or greater isolated left main stenosis.
* History of type 2 diabetes or metabolic syndrome at the time of study enrollment
* Willing to participate as evidence by signing the study informed consent

Exclusion Criteria:

1. Prior history of chronic infectious disease, including tuberculosis, severe fungal disease, or known HIV positive
2. Chronic hepatitis B or C infection
3. Interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis. Chest x-ray evidence in the past 12 months of interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis.
4. Prior history of non basal cell malignancy or myeloproliferative or lymphoproliferative disease within the past 5 years
5. White blood cell count <3,500/mm3, hematocrit <32%, or platelet count <75000/mm3
6. Liver transaminase levels (AST/ALT) greater than the upper limit of normal or albumin less than the lower limit of normal
7. Creatinine clearance (CrCl) <40 mL/min as estimated by the Cockcroft-Gault equation
8. History of alcohol abuse or unwillingness to limit alcohol consumption to <4 drinks per week
9. Women of child bearing potential, even if currently using contraception, and women intending to breastfeed
10. Men who plan to father children during the study period or who are unwilling to use contraception
11. Requirement for use of drugs that alter folate metabolism (trimethoprim/sulfamethoxazoyl) or reduce tubular excretion (probenecid) or known allergies to antibiotics making avoidance of trimethoprim impossible
12. Current indication for methotrexate therapy
13. Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers
14. Known chronic pericardial effusion, pleural effusion, or ascites
15. New York Heart Association class IV congestive heart failure
16. Life expectancy of <3 years

The study population for the ancillary study will be the same as the main trial with the following additional exclusion criteria

1. Subjects with a history of multiple imaging studies associated with radiation exposure
2. Insulin-dependent diabetics
3. If subject is Type 2 diabetic, hemoglobin A1c greater than 8% as determined by patient medical record review in the one year prior to the date of consent to this study.
4. BMI greater than 37 kg/m2 or weight greater than 350 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Fayad, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
- St. Michael's Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled period from Dec 2015 to April 2018
Groups:
- Low Dose Methotrexate: Low dose methotrexate - average dose of 15-20 mg po/weekly. will additionally receive 1 mg daily oral folate.
Period: Overall Study
Arm/Group | Low Dose Methotrexate | Placebo
Started | 60 | 63
Completed | 26 | 27
Not Completed | 34 | 36
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 11 | 0
Not completed — Withdrawal by Subject | 11 | 2
Not completed — study closure of main CIRT trial) | 0 | 8
Not completed — not randomized, failed run-in | 7 | 0
Not completed — screen failure/ re-enrolled | 0 | 25
Not completed — Physician Decision | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Methotrexate | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [61 to 67] | 65 [59 to 71] | 64 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 18 | 20 | 38
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
hs-CRP [Median (Inter-Quartile Range); unit: mg/L] | 1.4 [0.7 to 2.1] | 1.1 [0.7 to 2.1] | 1.3 [0.7 to 2.1]
Total Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 138.1 [108 to 160] | 131 [112 to 158] | 134 [108 to 160]
LDL cholesterol [Median (Full Range); unit: mg/dL] | 63 [49 to 84] | 66 [45.2 to 82] | 64 [45 to 84]
HDL cholesterol [Median (Full Range); unit: mg/dL] | 42.5 [38 to 50] | 40 [36.3 to 47] | 41.5 [36 to 50]
MDS TBR Index Vessel [Median (Inter-Quartile Range); unit: ratio] — Most Diseased Segment (MDS) Target to Background (TBR) Index Vessel
  ratio | 2.46 [2.15 to 2.77] | 2.41 [2.06 to 2.75] | 2.44 [2.06 to 2.77]
TMNMX MDS [Median (Full Range); unit: ratio] — TMNMX: TBR Mean of the Max MDS
  ratio
    LCC - left common carotid | 2.04 [1.89 to 2.29] | 2.12 [1.85 to 2.46] | 2.08 [1.85 to 2.46]
    RCC - right common carotid | 2.12 [2.04 to 2.48] | 2.13 [1.99 to 2.36] | 2.12 [1.99 to 2.48]
    ATA - ascending thoracic aorta | 2.45 [2.08 to 2.72] | 2.22 [1.97 to 2.71] | 2.34 [1.97 to 2.72]
TMNMX [Median (Inter-Quartile Range); unit: ratio] — TMNMX: TBR Mean of the Max
  ratio
    Combined Carotid | 1.93 [1.75 to 2.22] | 1.93 [1.77 to 2.24] | 1.93 [1.75 to 2.24]
    ATA | 2.34 [1.98 to 2.53] | 2.12 [1.92 to 2.58] | 2.23 [1.92 to 2.58]
SMNMX [Median (Full Range); unit: ratio] — Standardized uptake value mean of the maximum
  ratio
    Combined Carotid | 1.82 [1.63 to 2.20] | 1.78 [1.52 to 1.95] | 1.80 [1.52 to 2.20]
    ATA | 2.26 [1.95 to 2.53] | 2.24 [2.04 to 2.46] | 2.25 [1.95 to 2.53]

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Inflammation
Description: Change in arterial inflammation - The relative change at 8 months as compared to baseline in arterial inflammation as measured by the most diseased segment (MDS) of the index vessel. The MDS is defined as the 1.5 cm segment within the carotid artery (right or left carotid) that demonstrates the highest PET/CT activity, and is calculated as a mean of maximum TBR values derived from 3 contiguous axial segments. The index vessel in turn is defined as the vessel (either aorta, right, or left carotid) with the greatest mean TBR at baseline. (MDS TBR Index Vessel)
Time Frame: baseline and 8 months
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Low Dose Methotrexate | Placebo
Number analyzed (Participants) | 26 | 27
percent change | 0.03 [-0.19 to 0.30] | 0.20 [-0.06 to 0.42]

2. Secondary Outcome: Change in Max Target-to-background (TBR)
Description: Change in max target-to-background (TBR) - The mean of max TBR within the carotid arteries as an average of the slices from the left and right carotid) at follow up imaging as compared to baseline.
Time Frame: baseline and 8 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Low Dose Methotrexate | Placebo
Number analyzed (Participants) | 26 | 27
ratio | 0.06 [-0.08 to 0.21] | 0.02 [-0.20 to 0.15]

3. Secondary Outcome: Change in Max TBR Within the Carotid Arteries
Description: Change in max target-to-background (TBR) - The mean of max TBR within the carotid arteries as an average of the slices from the left and right carotid)
Time Frame: baseline and 8 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Low Dose Methotrexate | Placebo
Number analyzed (Participants) | 26 | 27
ratio | -0.04 [-0.29 to 0.12] | 0.06 [-0.14 to 0.20]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Low Dose Methotrexate | Placebo
All-Cause Mortality (participants affected / at risk) | 1/60 | 1/63
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 1/60 | 1/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Methotrexate (N=60) | Placebo (N=63)
Missinjected dose (isotope) (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT02576067/Prot_SAP_000.pdf